CLINICAL TRIAL: NCT06199401
Title: Safety and Efficacy of XJ-Procedure in Patients With Acute Type A Aortic Dissection Surgery (ADVANCED-XJ-Ⅱ): A National, Multi-center, Open-label, Randomized, Controlled, Blinded-end Point Trial
Brief Title: Safety and Efficacy of XJ-Procedure in Patients With Acute Type A Aortic Dissection Surgery
Acronym: ADVANCED-XJ-Ⅱ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Qinghai People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF2023LSYY-006-1
Record Dates: First submitted 2023-12-18; First posted 2024-01-10 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: Type A Aortic Dissection; Complication of Surgical Procedure; Aortic Diseases
Keywords: Type A Aortic Dissection; Aortic Root Reinforcement; Cardiovascular Surgery; Postoperative Complication
MeSH Terms: conditions — Aortic Diseases; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XJ-Procedure Group (Experimental): In the XJ-Procedure Group, Patients will be performed the standard "Sun's procedure" after general anesthesia, in which the end-to-end anastomosis between the artificial vessel and the aortic root is performed using the "Vascular Grafts Eversion and Built-in Technique" during the aortic root suture.
  Interventions: Procedure: Vascular Grafts Eversion and Built-in Technique(XJ-Procedure)
- Control Group (No Intervention): In the Control Group, Patients will be performed the standard "Sun's procedure" which involves aortic root anastomosis using the regular technique at each cardiovascular surgery center.

INTERVENTIONS:
Procedure: Vascular Grafts Eversion and Built-in Technique(XJ-Procedure) — A 1.5-2cm wide bovine pericardial patch and graft ring will be placed inside and outside the aortic root and against the aortic wall, respectively, and continuously sutured near the commissure using 5-0 polypropylene. Then an eversion about 15mm of vascular graft will be intermittently sutured to full layers of aortic vascular with 2-0 pad polyester suture. Finally, the eversion and aortic wall will be continuously sutured together in one more turn.
  Arms: XJ-Procedure Group

SUMMARY:
This is a national, multicenter, open-label, randomized, controlled, endpoint-blinded clinical trial of patients diagnosed with ATAAD and undergoing "Sun's procedure" coordinated by the First Affiliated Hospital of Xi'an Jiaotong University, China. Per the protocol, "Sun's procedure" combined with "XJ-Procedure" in the anastomosis of the aortic root and Sun's procedure combined with regular suturing methods of the aortic root will be compared.

DETAILED DESCRIPTION:
In this study, the investigators will prospectively enroll patients diagnosed with ATAAD and undergo "Sun's procedure" from November 2024 to November 2027 in several centers, including the First Affiliated Hospital of Xi'an Jiaotong University, and will randomly divide them into XJ-procedure group and control group. "The patients in the XJ-procedure group will undergo "Sun's procedure", in which the anastomosis of the aortic root will be performed with the XJ-procedure. The patients in the control group will also undergo "Sun's procedure", in which the anastomosis of the aortic root will be performed with each center. The primary outcome event is all-cause mortality within 12 months after surgery. Secondary outcome events are (1) incidence of residual aortic root entrapment (during hospitalization, follow-up 3 months, 6 months, 12 months) (2) rate of secondary surgery for hemostasis due to root hemorrhage (during hospitalization) (3) incidence of anastomotic pseudoaneurysm (during hospitalization, follow-up 3 months, 6 months, 12 months) (4) rate of severe regurgitation of residual aortic valves (during hospitalization, follow-up 3 months, 6 months, 12 months) (5) Incidence of major adverse cardiovascular and cerebrovascular events (MACCE) (during hospitalization, follow-up 3 months, 6 months, 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years;
* Patients with ATAAD attending the relevant department who have been assessed by a clinician as needing "Sun's procedure".

Exclusion Criteria:

* Severe aortic root involvement (root diameter >45 mm, root tear, severe destruction of the aortic root, combined valve disease);
* Combined coronary artery disease requiring concomitant coronary revascularization;
* Prior aortic or cardiac surgery;
* Preoperative severe malperfusion syndromes such as: severe cerebral complications (acute cerebral infarction, cerebral hemorrhage, coma, etc.); malperfusion of abdominal organs or lower extremities >12 h;
* Preoperative combination of severe single or multiple organ failure;
* Pregnant women;
* Refused to sign the informed consent form and refused to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months follow-up
  This outcome is a time-to-event variable and its data will be obtained at 12 months follow-up, according to the medical records or phone calls of all patients.

SECONDARY OUTCOMES:
Change of incidence of residual aortic root dissection | About 20 days (during hospitalization), at the 3 months, 6 months, and 12 months follow-up
  The data will be obtained during hospitalization, at the 3 months, 6 months, and 12 months follow-up, according to CTA and echocardiography results of all patients.
Change of incidence of second surgery for hemostasis due to aortic root hemorrhage | About 20 days (during hospitalization)
  The data will be obtained during hospitalization, according to medical records of all patients.
Change of incidence of anastomotic pseudoaneurysms during hospitalization | About 20 days (during hospitalization), at the 3 months, 6 months, and 12 months follow-up
  The data will be obtained during hospitalization at the 3 months, 6 months, and 12 months follow-up, according to CTA and echocardiography results of all patients.
Change of incidence of severe residual aortic valve regurgitation | About 20 days (during hospitalization), at the 3 months, 6 months, and 12 months follow-up
  The data will be obtained during hospitalization, at the 3 months, 6 months, and 12 months follow-up, according to the echocardiography results of all patients.
Change of incidence of MACCE | About 20 days (during hospitalization), at the 3 months,6 months, and 12 months follow-up
  MACCE includes all-cause of death, myocardial infarction, stroke and coronary revascularization. The data will be obtained during hospitalization, at the 3 months, 6 months, and 12 months follow-up, according to medical records and imaging findings of all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China